CLINICAL TRIAL: NCT03857971
Title: Identification of Risk Factors for Acute Coronary Events by Optical Coherence Tomography After STEMI and NSTEMI in Patients With Residual Non-flow Limiting Lesions The 'PECTUS-obs' Trial (Observational Cohort)
Brief Title: Identification of Risk Factors for Acute Coronary Events by OCT After STEMI and NSTEMI in Patients With Residual Non-flow Limiting Lesions
Acronym: PECTUS-obs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NL67426.091.18
Record Dates: First submitted 2019-02-27; First posted 2019-02-28 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease
Keywords: Vulnerable plaque; Optical coherence Tomography; OCT
MeSH Terms: conditions — Myocardial Infarction; Acute Coronary Syndrome; Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronary OCT imaging of non flow-limiting lesion (Other): Coronary OCT imaging will be performed of fractional flow reserve (FFR) negative lesions to assess plaque morphology.
  Interventions: Device: Coronary Optical Coherence tomography

INTERVENTIONS:
Device: Coronary Optical Coherence tomography — Optical coherence tomography imaging is performed of non-obstructive, non-culprit coronary lesions to assess plaque morphology.

SUMMARY:
The objective of this study is to compare the clinical outcome of Non-ST-elevation myocardial infarction (NSTEMI) and ST-elevation myocardial infarction (STEMI) patients with non-obstructive, non-culprit coronary lesions and either presence or absence of vulnerable plaque characteristics as assessed by optical coherence tomography (OCT).

DETAILED DESCRIPTION:
Despite major advances in the treatment of acute coronary syndromes a large proportion of patients is still at risk for new coronary events after experiencing an acute coronary syndrome (ACS). Detection of residual vulnerable plaques after ACS using OCT potentially identifies patients at high risk for new coronary events. However, no prospectively collected data on the prognostic power of OCT for plaque rupture are available at this moment. To design trials aimed to reduce events in patients with vulnerable plaques it is required to collect such prospective data on the relation between OCT derived characteristics of vulnerability and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent must be obtained.
* Patients with STEMI or NSTEMI and residual, non-culprit CAD, with the possibility of plaque vulnerability.
* Residual plaque(s) is(are) non-obstructive (FFR≥0.80).

Exclusion Criteria:

* Refusal or inability to provide informed consent.
* < 18 years of age
* Hemodynamic instability, respiratory failure, Kilip class ≥ 3.
* Previous Coronary Artery Bypass Grafting (CABG).
* Indication for revascularization by CABG.
* Anatomy or lesions unsuitable for OCT catheter crossing or imaging (aorta-ostial lesions, small diameter segment, severe calcifications, lesion is too distal for OCT catheter)
* Pregnancy.
* Estimated life expectancy < 3 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2018-12-14 (Actual); Primary Completion 2022-09-15 (Estimated); Study Completion 2025-06-14 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac Events | 2 years
  Composite of all cause mortality, non-fatal myocardial infarction or unplanned revascularization.

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 1 year
  Composite of all cause mortality, non-fatal myocardial infarction or unplanned revascularization.
Major Adverse Cardiac Events | 5 years
  Composite of all cause mortality, non-fatal myocardial infarction or unplanned revascularization.
Target lesion Failure | 2 and 5 years
  Cardiac death caused by target lesion, myocardial infarction caused by target lesion, revascularisation of target lesion

CONTACTS AND LOCATIONS:
Overall Officials: Niels van Royen, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Volleberg RHJA, Rroku A, Mol JQ, Hermanides RS, van Leeuwen M, Berta B, Meuwissen M, Alfonso F, Wojakowski W, Belkacemi A, Roleder T, Kedhi E, van Royen N; COMBINE (OCT-FFR) and PECTUS-obs investigators. FFR-Negative Nonculprit High-Risk Plaques and Clinical Outcomes in High-Risk Populations: An Individual Patient-Data Pooled Analysis From COMBINE (OCT-FFR) and PECTUS-obs. Circ Cardiovasc Interv. 2025 Feb;18(2):e014667. doi: 10.1161/CIRCINTERVENTIONS.124.014667. Epub 2025 Jan 22. PMID 39840429
- [Derived] Volleberg RHJA, Mol JQ, Belkacemi A, Hermanides RS, Meuwissen M, Protopopov AV, Laanmets P, Krestyaninov OV, Lacle CF, Oemrawsingh RM, van Kuijk JP, Arkenbout K, van der Heijden DJ, Rasoul S, Lipsic E, Rodwell L, Camaro C, Damman P, Roleder T, Kedhi E, van Leeuwen MAH, van Geuns RM, van Royen N. High-risk plaques in non-culprit lesions and clinical outcome after NSTEMI vs. STEMI. Eur Heart J Cardiovasc Imaging. 2025 Jan 31;26(2):197-206. doi: 10.1093/ehjci/jeae289. PMID 39512201
- [Derived] Mol JQ, Belkacemi A, Volleberg RH, Meuwissen M, Protopopov AV, Laanmets P, Krestyaninov OV, Dennert R, Oemrawsingh RM, van Kuijk JP, Arkenbout K, van der Heijden DJ, Rasoul S, Lipsic E, Teerenstra S, Camaro C, Damman P, van Leeuwen MA, van Geuns RJ, van Royen N. Identification of anatomic risk factors for acute coronary events by optical coherence tomography in patients with myocardial infarction and residual nonflow limiting lesions: rationale and design of the PECTUS-obs study. BMJ Open. 2021 Jul 7;11(7):e048994. doi: 10.1136/bmjopen-2021-048994. PMID 34233996